CLINICAL TRIAL: NCT06162871
Title: The Effect of Social Participation As a Key Determinant of Healthy Aging
Brief Title: Social Participation and Healthy Aging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Collaborators: Fondazione Sardegna (Unknown)
Responsible Party: Principal Investigator, Giulia Cossu, Principal Investigator, University of Cagliari
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NP.2023/2534
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy Aging
Keywords: healthy aging; Generational exchange; Psychosocial intervention; Pilot study

STUDY DESIGN:
Intervention Model Description: The experimental condition in the experimental group consists of a psychosocial intervention. The control group is initially inactive and after the experimental group post treatment will be involved in the experimental intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active participation (Experimental)
  Interventions: Behavioral: Presentations and interactive debate sessions, with intergenerational exchange
- non involved in active part (No Intervention)

INTERVENTIONS:
Behavioral: Presentations and interactive debate sessions, with intergenerational exchange — Intervention will consist of 12 sessions, each lasting about two hours, conducted on a weekly basis and delivered both in-person and remotely. The sessions will include presentations and interactive debate sessions, with a central focus on intergenerational exchange covering cultural, historical, and health-related topics. A key aspect is the active involvement of beneficiaries, individuals over sixty-five, who will be asked to prepare presentations with the support of project-provided facilitators. Simultaneously, the project will promote and enhance skills, organizational capabilities, and computer literacy.
  Arms: active participation

SUMMARY:
The research aims to promote active aging through a pilot study. The design will be crossover with two groups. Intervention will consist of presentations and interactive debate sessions, with a central focus on intergenerational exchange covering cultural, historical, and health-related topics. A key aspect is the active involvement of beneficiaries, individuals over sixty-five. The outcomes will be quality of life, presence of depressive symptoms, and regularity of biological and social rhythms.

DETAILED DESCRIPTION:
In 2050, 36% of the Italian population will be over 65 years old. The European Union has identified as a priority the increase in research on active aging, promoting activities that can maintain and enhance the health and social engagement of individuals aged 65 and above.

This pilot study aims to assess feasibility a preliminary measure of effectiveness of a psychosocial intervention focused on intergenerational exchange on quality of life, biological and social rhythms, and mood in a group of elderly

The outcomes will include quality of life, presence of depressive symptoms, and regularity of biological and social rhythms, assessed before the intervention, immediately after intervention and at a follow-up four months after the intervention's conclusion.

The psychosocial intervention will consist of sessions on a weekly basis and delivered both in-person and remotely. The sessions will include presentations and interactive debate sessions, with a central focus on intergenerational exchange covering cultural, historical, and health-related topics. A key aspect is the active involvement of beneficiaries, individuals over sixty-five, who will be asked to prepare presentations with the support of project-provided facilitators. Simultaneously, the project will promote social inclusion, enhance skills, organizational capabilities, and computer literacy.

ELIGIBILITY:
Inclusion Criteria:

* people who are 65 years of age or older

Exclusion Criteria:

* have serious problems with independent walking,
* have serious neurological conditions or serious disabilities that make it impossible to participate in the intervention in person or remotely

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to post treatment and to follow-up of The Short Form Health Survey (Quality of life) | T0 (0 weeks); T1 (12 weeks); T2 (28 weeks)
  To evaluate it will be used: The Short Form Health Survey (SF-12), a brief version of SF-36 questionnaire, made up of twelve questions, values range from 12 to 47, includes the following dimensions: physical activity, disturbance in physical health, physical condition, self-assessment of health status, vitality, social activity and mental health assessed on a monthly basis . Higher scores recorded a greeting and better Quality of life
Change from Baseline to post treatment and to follow-up of The Brief Social Rhythms Scale (Social and biological Rhythms) | T0 (0 weeks); T1 (12 weeks); T2 (28 weeks)
  To evaluate it will be used: The Brief Social Rhythms Scale (BSRS), a 10 item questionnaire, values range from 10 to 60, designed to assess the level of regularity in biological and social rhythms, specifically those related to sleep-wake cycles and appetite, as well as social contacts. Higher scores recorded a worse regulation of rhythms
Change from Baseline to post treatment and to follow-up of Patient Health Questionnaire-9 (Depression symptoms) | T0 (0 weeks); T1 (12 weeks); T2 (28 weeks)
  To evaluate it will be used: Patient Health Questionnaire-9 (PHQ-9) a short self-administered tool, values range from 0 to 27, used for screening, diagnosis, monitoring and measuring the severity of depression. It's composed of 9 items that correspond to the symptoms of major depression according to DSM-IV on last two weeks. Higher scores identify a greater presence of depressive symptoms.
Change from Baseline to post treatment and to follow-up of Physical Activity Questionnaire (type and quantity of physical activity) | T0 (0 weeks); T1 (12 weeks); T2 (28 weeks)
  To evaluate it will be used: Physical Activity Questionnaire (IPAQ) designed to measure the type and quantity of physical activity undertaken in the past 7 days, values range from 0 to the maximum amount of minutes a person spends on physical activity or sedentary activities, including occupational and recreational physical activities, through 9 items, on a weekly basis, Higher scores identify in a subscale a frequent physical activity (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Change from Baseline to post treatment and to follow-up of Addenbrooke's Cognitive Examination (Cognitive performance) | T0 (0 weeks); T1 (12 weeks); T2 (28 weeks)
  To evaluate it will be used: Addenbrooke's Cognitive Examination (ACE-R), a brief cognitive test, values range from 0 to 100, that assesses five cognitive areas: attention/orientation, memory, verbal fluency, language, and visuo-spatial abilities. The test incorporates the Mini Mental State Examination (MMSE).
  The higher the score obtained in the test, the lower the presence of signs that identify cognitive deterioration on the screening performance scales
Evaluation of the Feasibility of the intervention with Dropout rate at post intervention time | at T1 (12 weeks)
  To evaluate it will be used: Dropout rate (25% dropout in the sample will be considered acceptable considering that it is a group of elderly people)
Intervention satisfaction at post intervention time | at T1 (12 weeks)
  Intervention satisfaction questionnaire (it will be considered a satisfactory level if on average the intervention is rated by the participants one standard deviation above the average of the ad hoc questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni di Dio Hospital, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cossu G, Lorrai S, Galetti A, Perra A, Tusconi M, Carra G, Preti A, Holzinger A, Carta MG. Promoting healthy aging through intergenerational exchange and digital empowerment: a pilot randomized controlled trial. Front Psychiatry. 2025 Jul 16;16:1637181. doi: 10.3389/fpsyt.2025.1637181. eCollection 2025. PMID 40740264